CLINICAL TRIAL: NCT05178875
Title: Estimation of Dietary and Urinary Nitrate Concentration in a Representative UK Population Using Data From the National Diet and Nutrition Survey (Years 1-8).
Brief Title: Estimation of Dietary Nitrate Intake in a Representative UK cohort_V1
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, prof, University of Reading
Other Study IDs: 18/NS/0085
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Nitrate Vasodilator Adverse Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NDNS participants: Random participants from all the UK (including England, Scotland, Wales and North Ireland)

SUMMARY:
Dietary nitrate has been shown to have health benefits including lowering blood pressure and improving the health and elasticity of blood vessels. The main source of dietary nitrate in the human diet is vegetables. Drinking water is another important contributor to nitrate intake but the nitrate level of drinking water varies on a daily basis and between different water authorities in the UK. Furthermore, the data available on dietary analysis software on the levels of nitrate in vegetables and vegetable-based foods is very limited. Therefore, there is an urgent need to more accurately estimate the levels of dietary nitrate intake in the UK population, and determine how the level of intake from all dietary sources (vegetables and drinking water) relate to risk factors for developing heart disease.

This project aims to analyse biobanked urine samples collected during Years 1 to 8 of the National Diet and Nutrition Survey (NDNS), which is conducted in a representative sample of the UK population. We will measure the levels of nitrate and its break down products (metabolites) in urine by using HPLC to estimate the levels of intake of dietary nitrate in the study participants. In addition, we will determine the level of intake from the diet diaries of the study participants using our database of nitrate levels in vegetables and drinking water to estimate the dietary intake, and compare this data with the urine analysis as a potential biomarker of dietary intake.

The NDNS study participants have previously consented for their urine samples to be used for future tests relating to nutrition and health as long as these tests have been approved by a NHS ethics committee. We have been granted permission to analyse the urine samples by the NDNS Bioresource Panel but must first gain ethical approval before the samples can be released to us for

DETAILED DESCRIPTION:
In this laboratory study, we will estimate the average dietary nitrate intake of each participant of the NDNS study using both the analyse of 2500 biobanked urine samples collected from participants of the National Diet and Nutrition Survey. As part of the consent process for the 24 h urine collection for the NDNS study (NREC reference number 07/H0604/113) participants were given the option to consent for any of their remaining urine samples to be used in tests relating to nutrition and health which had been approved by a NHS ethics committee.

The main inclusion criteria of this laboratory project are:

- Adults aged 19-64 y with a complete 4-day diet diary and a biobanked urine sample

For the dietary analysis, the nitrate levels of each food item consumed (mainly vegetables and drinking water) will be estimated using UK and European food nitrate values and from previously published studies in the literature. In addition, the nitrate content of drinking water will be estimated for each participant by contacting DWI and the local water suppliers in the UK to collect the quality control of the nitrate content of the drinking water in the UK. The nitrate and nitrite level data will be sent to the NatCen Social Research staff to match the data to each participant based on their postcode and the year the volunteers participated in the NDNS study.

To associate the estimated daily intake of dietary nitrate with health markers and risk factors for cardiovascular disease, analysis of covariance will be used to detect statistically significant differences between high and low nitrate containing diets with blood pressure and other risk factors for cardiovascular disease, controlling for age, sex and total energy intake (MJ). Post-hoc pair-wise analysis will detect differences between quartiles of dietary nitrate intake.

To compare the agreement of the urine nitrate data with the dietary nitrate data, statistical tests such as Bland Altman analysis and principal components analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19-64 y with a complete 4-day diet diary and a biobanked urine sample

Exclusion Criteria:

* not consented to the future analysis of the biobanked urine sample for nutrition and health research
* the diet diary was not completed
* insufficient urine sample available for the urinary nitrate and metabolite analysis.

Ages: 19 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Healthy participants
Sampling Method: Probability Sample
Enrollment: 2444 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
The relationship between the estimated daily dietary nitrate intake with blood pressure and other risk factors for cardiovascular disease in UK adults (aged 19-64 years) of the National Diet and Nutrition Survey. | 1 year
  The daily nitrate intake will be estimated from both analysis of urine samples for nitrate and its metabolites, and also from the diet diary.

SECONDARY OUTCOMES:
associations between diets containing high and low intakes of nitrate with blood pressure and other risk factors for cardiovascular disease | 1 year
  participant will be devided in quartiles based on their nitrate intake then link these data with blood pressure and other CVD risk factors.
if measurement of nitrate and its metabolites in urine represents a suitable biomarker to estimate dietary nitrate intake. | 1 year
  urinary nitrate will be compared with nitrate intake and linked with blood pressure and other CVD risk factors and

CONTACTS AND LOCATIONS:
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alzahrani HS, McKenna HB, Hobbs DA, Jackson KG, Lovegrove JA. Dietary Sources of Nitrate and Nitrite and Associations with Blood Pressure and Other Cardiovascular Disease Risk Factors in a Representative United Kingdom Population. J Nutr. 2025 Nov 24:101249. doi: 10.1016/j.tjnut.2025.11.018. Online ahead of print. PMID 41297631